CLINICAL TRIAL: NCT05487898
Title: Benefits of Cycling Wheelchair Training for Elderly With Physical Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CE22294A
Record Dates: First submitted 2022-06-19; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-06

CONDITIONS: Aged; Disable; Exercise; Rehabilitation; Wheelchair
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cycyling wheelchair (Experimental): Volunteers join the cycling wheelchair training
  Interventions: Device: Cycling wheelchair

INTERVENTIONS:
Device: Cycling wheelchair — Apply the mechanical principle of pedaling on a bicycle to a conventional wheelchair

SUMMARY:
To investigate the feasibility of cycling wheelchair training as an exercise for elderly disabled patients, and to determine its effects on cognition, quality of life, aerobic capacity and physiological markers. We measure SF-12. Other outcome measures included the Mini-Mental State Examination, Aero bike workload test, resting blood pressure (systolic and diastolic), and heart rate.

ELIGIBILITY:
Inclusion Criteria:

1. age >65 years old
2. with a functional ambulation category scale (FAC) level 4 or below
3. muscle strength of both lower limbs was >3 as the , or the muscle strength of one lower limb was 4 or above, as rated by the Medical Research Council Scale (MRC).

Exclusion Criteria:

1. hospitalized for acute medical problems within the past 3 months
2. having cardiopulmonary disease that could cause exercise hazards
3. unable to perform repetitive pedaling exercise due to diseases of the lower limbs
4. with pressure ulcers around hip area
5. with impaired cognitive function that did not allow completion of our questionnaires.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
SF-12 | one month
  Quality of life
MMSE questionnaire | one month
  Cognitive function
Cycling ergometer | one month
  Aerobic capacity

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No discuss with volunteers about sharing data to third party

REFERENCES:
- [Derived] Fu JC, Fu PK, Cheng YY. Benefits of Cycling Wheelchair Training for Elderly with Physical Disability: A Prospective Cohort Study. Int J Environ Res Public Health. 2022 Dec 14;19(24):16773. doi: 10.3390/ijerph192416773. PMID 36554652